CLINICAL TRIAL: NCT04271514
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-dose Escalation, Multiple-dose Escalation, and Food Effect Study of RPT193 in Healthy Subjects and Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A First-in-Human Study of RPT193 in Healthy Volunteers and Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPT193-01
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- COMPLETED ENROLLMENT -- Single Dose Escalation Part A - active (Experimental): Increasing doses of RPT193 will be administered to healthy volunteers
  Interventions: Drug: RPT193
- COMPLETED ENROLLMENT -- Single Dose Escalation Part A - placebo (Placebo Comparator): Matching placebo will be administered to healthy volunteers
  Interventions: Drug: Placebo
- COMPLETED ENROLLMENT -- Multiple Dose Escalation Part B - active (Experimental): Increasing doses of RPT193 will be administered once/day for 7 days to healthy volunteers
  Interventions: Drug: RPT193
- COMPLETED ENROLLMENT -- Multiple Dose Escalation Part B - placebo (Placebo Comparator): Matching placebo will be administered once/day for 7 days to healthy volunteers
  Interventions: Drug: Placebo
- COMPLETED ENROLLMENT -- Expansion Part C - active (Experimental): RPT193 will be administered daily for 28 days to patients with atopic dermatitis
  Interventions: Drug: RPT193
- COMPLETED ENROLLMENT -- Expansion Part C - placebo (Placebo Comparator): Matching placebo will be administered daily for 28 days to patients with atopic dermatitis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPT193 — Antagonist of the CCR4 chemokine receptor
  Arms: COMPLETED ENROLLMENT -- Expansion Part C - active; COMPLETED ENROLLMENT -- Multiple Dose Escalation Part B - active; COMPLETED ENROLLMENT -- Single Dose Escalation Part A - active
Drug: Placebo — Matching placebo
  Arms: COMPLETED ENROLLMENT -- Expansion Part C - placebo; COMPLETED ENROLLMENT -- Multiple Dose Escalation Part B - placebo; COMPLETED ENROLLMENT -- Single Dose Escalation Part A - placebo

SUMMARY:
This study is a first-in-human, 3-part, multi-center, Phase 1, randomized, double-blind, placebo-controlled study with RPT193 in up to 64 healthy male and female subjects and 30 male and female patients with atopic dermatitis. RPT193 is an orally-available, potent, and selective antagonist of CCR4.

ELIGIBILITY:
Selected Inclusion Criteria:

Parts A & B (COMPLETED ENROLLMENT):

* Healthy male or female
* 18-55 years of age, inclusive
* At least 50 kg in weight
* BMI: 18.0-30.0 kg/m2, inclusive

Part C (COMPLETED ENROLLMENT):

* Male or female with atopic dermatitis
* 18-65 years of age, inclusive
* BMI between 18.0 (inclusive) and <40.0 kg/m2
* Body surface area (BSA) with AD involvement ≥10%
* Eczema Area and Severity Index (EASI) score ≥12
* Validated Investigator's Global Assessment (vIGA) ≥3
* History of inadequate response to treatment with topical medications, such as corticosteroids or calcineurin inhibitors, or patients for whom topical treatments are otherwise medically inadvisable

Selected Exclusion Criteria:

Parts A & B (COMPLETED ENROLLMENT):

* Use of tobacco products within 60 days prior to drug administration
* History of alcohol abuse or drug addiction
* Positive drug and alcohol screen
* Participation in a drug study within 60 days prior to drug administration
* Donation or loss of more than 100 mL of blood within 60 days prior to drug administration.
* Donation or loss of more than 1.5 liters of blood (for male subjects) / more than 1.0 liters of blood (for female subjects) in the 10 months prior to drug administration.

Part C (COMPLETED ENROLLMENT):

* Any serious and/or uncontrolled medical condition
* History of alcohol abuse or drug addiction
* Positive drug and alcohol screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | up to Day 16 (Part A: SAD); up to Day 22 (Part B: MAD); up to Day 43 (Part C)
  Number of participants with abnormal laboratory values and/or adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Cheng, MD, PhD, Study Director — RAPT Therepeutics, Inc.
Locations (14):
- United States (13):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Perseverance Research Center LLC, Scottsdale, Arizona
  - University Clinical Trials, Inc, San Diego, California
  - Lenus Research & Medical Group, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Clinical Trials Management,LLC, Metairie, Louisiana
  - MetroBoston Clinical Partners LLC, Brighton, Massachusetts
  - Sadick Research Group LLC, New York, New York
  - Central Sooner Research, Norman, Oklahoma
  - DermResearch, Inc., Austin, Texas
  - Progressive Clinical Research PA, San Antonio, Texas
- PRA, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No